CLINICAL TRIAL: NCT06966323
Title: Hold me Tight/Let me Go: Effectiveness of a Course to Enhance Parent-adolescent Relationship
Status: Recruiting | Type: Observational
Sponsor: University of Amsterdam (Other)
Responsible Party: Principal Investigator, Henk Jan Conradi, Assistant Professor of Clinical Psychology, University of Amsterdam
Other Study IDs: FMG-12034
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Parent Training; Parent Child Relationship; Parent-child Problem
Keywords: Hold Me Tight Program; Emotionally Focused Therapy; Parent Child Problems; Parent Child Relationships; Adolescents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Hold me Tight / Let me Go — Hold Me Tight / Let Me Go (HmT/LmG) is a manualized, group-based behavioral intervention for parents of adolescents aged 12 to 18. Grounded in Emotionally Focused Therapy (EFT) and Hold me Tight for couples. HmT/LmG aims to improve the parent-adolescent relationship by enhancing emotional validation, secure attachment, and effective communication.
  The intervention consists of four group sessions for parents, supplemented by three structured individual or dyadic sessions involving both parents and adolescents. Key components include psycho-education, role plays, emotion-focused conversations, and exercises targeting validation, apologizing, and supportive limit setting. Families complete pre- and post-intervention questionnaires and a follow-up assessment to evaluate changes in relationship quality and psychological well-being.

SUMMARY:
HmT/LmG is a group course for 4-6 parental dyads and consists of 4 group sessions with psycho-education and skills training and 3 individual sessions per family (i.e., 1 session with the adolescent, 1 session with the parents, and 1 session with parents and adolescent together). We want to evaluate effectiveness and treatment process mechanisms applying self-reports, audio observation and interviews.

DETAILED DESCRIPTION:
HOLD ME TIGHT/LET ME GO: STUDY PROTOCOL (version 2025-05-01) Participants In- and exclusion criteria will be determined with unstructured clinical interviews by experienced clinicians during the screening.

Inclusion criteria:

1. Families with one or both parents/primary caretaker (single parent or blended families are allowed) with one adolescent of 12 to 18 years of age;
2. Adolescent problems are deemed to be exacerbated by a stressful parent-adolescent relationship.

Exclusion criteria:

1. Participants in command of the Dutch language.
2. Parents/primary caretakers and adolescents with severe psychopathology (e.g., psychosis, acute suicidality, severe depression) that will interfere with participation in the program.
3. Parents/primary caretakers already attending systemic therapy or intensive parental guidance during the waiting period and during HmT/LmG. Other individual therapy will be registered during intake, and afterwards by the therapists. During follow-up systemic interventions are allowed but have to be registered.

Design A randomized design comparing the intervention with a control group is not deemed feasible as this requires the simultaneous consent of families (i.e., father, mother and adolescent) to be randomized, which is much harder to achieve than with individuals. Further, the group format of the program (4 to 6 families) requires randomization of 8 to 12 families to be completed within a reasonable time frame otherwise families that were first randomized may drop out. From earlier experiences with randomization of groups of couples is known that this is not feasible because it will compromise inclusion unacceptably. Moreover, it was concluded that studies aiming at relationship enhancement may not need to include waitlist control groups as two meta-analyses found no statistically significant spontaneous improvement from relational problems (Baucom et al., 2003; Roddy et al., 2020). This is in contrast with depression which is known for its high spontaneous remission rates.

All in all, a within-subjects design will be used in which families serve as their own controls with three waves: waiting-period, treatment and follow-up. The waiting period will span on average five weeks (i.e., two to eight weeks), the treatment phase will last about 6 weeks, followed by a follow-up period of about 8 weeks). Change across the three waves will be compared. Little change is anticipated little change during the waiting period (indicating no spontaneous remission), gain during treatment, and little change (substantial maintenance) during follow-up.

Hypotheses:

1. ∆ waiting period < ∆ intervention period
2. M post-intervention period ≈ M follow-up period To enable these comparisons all questionnaires must be administered at least four times (pre-waiting, pre-treatment, post-treatment, follow-up)

Procedure: intervention and assessments

The intervention is a course for groups of parents from 4-6 families to help them to enhance their relationship with their adolescent child. The procedure plus timeline for parents and adolescents will be:

1. Parents intake session (8 to 2 weeks prior to session 1, duration 45-60 min.) is part of the standard procedure of the participating clinical practice.

   Goal: determining whether parents and adolescent are eligible for the HmT/LmG program.

   Measurements: (a) parents: paper and pencil (14 min., see measurement scheme parents), and (b) adolescent: paper and pencil when coming along with the parents otherwise via Qualtrics (11 min., see measurement scheme adolescents).
2. Parents group session 1 (2 to 8 weeks after intake, duration 150 min.). Goal: parents receive psycho-education about: (a) basic adolescent's needs (safe bonding with parents, validation, and autonomy to discover their identity), (b) the importance of parents being open and helpful (the building blocks of secure attachment) to facilitate fulfillment of the adolescent's needs, and (c) recognition of negative parent-adolescent interaction patterns that thwart need fulfillment. Exercises and role play on recognition of negative patterns and their effects are included.

   Measurement: (a) parents: paper and pencil (14 min.), and (b) adolescent: Qualtrics (11 min.).
3. Parents group session 2 (1 week after session 1, duration: 150 min.). Goal: parents receive psycho-education about: (a) self-protective behavior modes that underlie the negative interaction pattern, (b) attachment underlying self-protective behavior, (c) how to de-escalate and validate their adolescent. Exercises and role play on validation are included.

   Measurement: (a) parents: paper & pencil (5 min.).
4. Parents group session 3 (2 weeks after session 2, duration: 150 min.). Goal: parents receive psycho-education about: (a) stop escalation and start being open and helpful, (b) apologizing when the negative patterns re-emerges, ad (c) limit-setting to their adolescent. Exercises and role play on apologizing and limit setting are included.

   Measurements: (a) parents: paper & pencil (6 min.).
5. Adolescent individual session (between group sessions 3 and 4, duration: 30-45 min.).

   Goal: adolescent interviewed by EFT therapist about: (a) negative patterns with the parents, and (b) unfulfilled needs.

   Measurement: (a) adolescent: live Qualtrics (8 min.). PhD student will take care of this.
6. Parents individual session (between group sessions 3 and 4, duration: 90 minutes).

   Goal: parents are prepared by an EFT therapist to a conversation with their adolescent aiming at restoring: (a) staying open and helpful, (b) help their adolescent to fulfil their needs, (c) without relapsing into the negative pattern.

   Measurement: parents: paper & pencil (6.5 min.).
7. Parents-adolescent individual session (between sessions 3 and 4, duration: 90 min.).

   Goal: restoring the secure bond with parents and adolescents refraining from the negative pattern, and the adolescent is stimulated to be open about his/her unfulfilled needs, while the parents have to stay open & helpful to the adolescents needs (i.e., repairing the secure bond by the three learned skills apologizing, validating and safe limit setting) Measurements: parents: paper & pencil (6 min.), and (b) adolescent: paper & pencil (7 min.), and EFT therapist: (c) audio recording of the session, and (d) scoring the degree of goal attainment for this sessions.
8. Parents group session 4 (3 weeks after session 3, duration: 150 min.). Goal: parents receive psycho-education about: (a) summary of the core content of the course. Exercises and role play on (aspects) of restoring the secure bond, and reading emotions and facilitation of needs of the adolescent.

   Measurements: (a) parents: paper & pencil (12 min.), and (b) adolescent: Qualtrics (11 min.).
9. Parents-adolescent follow-up interview (8 weeks after session 4, duration 30-60 min.).

Goal: interview with parent(s) and adolescent about working mechanisms of HmT/LmG, testing a (initial) program theory (realist evaluation) to identify causal processes by examining how the program outcomes are caused by which underlying mechanisms within specific contexts.

Measurements: parents: live Qualtrics (12 min.), and (b) adolescent: live Qualtrics (11 min.), and (c) parents and adolescent: record of live qualitative interview via Zoom (30-60 min.).

ELIGIBILITY:
We will include:

1. Families with one or both parents/primary caretaker (single parent or blended families are allowed) with one adolescent of 12 to 18 years of age;
2. Adolescent problems are deemed to be exacerbated by a stressful parent-adolescent relationship.

We will exclude:

1. Participants in command of the Dutch language.
2. Parents/primary caretakers and adolescents with severe psychopathology (e.g., psychosis, acute suicidality, severe depression) that will interfere with participation in the program.
3. Parents/primary caretakers already attending systemic therapy or intensive parental guidance during the waiting period and during HmT/LmG. Other individual therapy will be registered during intake, and afterwards by the therapists. During follow-up systemic interventions are allowed but have to be registered.

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Families with adolescents aged 12 to 18 years will be recruited via participating clinical practices (mental health organizations) in the Netherlands. Recruitment will focus on families experiencing difficulties in the parent-adolescent relationship that are believed to contribute to the adolescent's emotional or behavioral problems. The population includes single-parent families, two-parent families, and blended families. The intervention is offered in the context of regular care.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in relationship satisfaction (CSI-4) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Positive change in relationship satisfaction of partners and adolescents (partners will report about their partner relationship, and parents and adolescents report about the parent-adolescent relationship). Satisfaction with the partner relationship of the parents, and the parent-adolescent relationship will be assessed with the 4 item Couple Satisfaction Index (CSI-4; Funk & Rogge, 2007).
  Funk, J. L., & Rogge, R. D. (2007). Testing the ruler with item response theory: Increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. Journal of Family Psychology, 21(4), 572-583. https://doi.org/10.1037/0893-3200.21.4.572
Change in negative patterns (RDS) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Negative change in negative patterns of partners and parents (partners will report about their partner relationship and parents and adolescents report about the parent-adolescent relationship). Negative patterns between the parents as partners and between parents and adolescent will be measured by the Relationship Dynamics Scale (RDS; Stanley et al., 2006) a four item self-report questionnaire. An example item is: 'When we argue, one of us withdraws, that is, does not want to talk about it anymore or leaves the scene.'
  Stanley, S. M., Amato, P. R., Johnson, C. A., & Markman, H. J. (2006). Premarital education, marital quality, and marital stability: Findings from a large, random household survey. Journal of Family Psychology, 20(1), 117-126. https://doi.org/10.1037/0893-3200.20.1.117

SECONDARY OUTCOMES:
Adolescents psychological need fulfillment (BPNS-9) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Increase in psychological need fulfillment of adolescents (adolescents will report about themselves). Need fulfillment in the context of the parent-adolescent relationships will be measured with the 9 item Basic Psychological Need Satisfaction in Relationships scale (BPNS-R). The adolescent version is based on the partner version (La Guardia, Ryan, Couchman, & Deci, 2000) and inspired in its wording by the Flemish version (Van der Kaap-Deeder et., 2020).
  La Guardia, J. G., Ryan, R. M., Couchman, C. E., & Deci, E. L. (2000). Within-person variation in security of attachment: A self-determination theory perspective on attachment, need fulfillment, and well-being. Journal of Personality and Social Psychology, 79, 367-384. http://doi.org/dhghf4
  Van der Kaap-Deeder, J., Soenens, B., Ryan, R. M., & Vansteenkiste, M. (2020). Manual of the Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS). Ghent University, Belgium.
Adolescents support seeking to parent (IERQ-3) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Increase in support seeking behavior of partners and adolescents (parents will report about their partner relationship and adolescents about the parent-adolescent relationship). Support seeking will be measured with a slightly adapted version of the Soothing subscale of the Interpersonal Emotion Regulation Questionnaire (IERQ; Hofman et al., 2016). We shortened the original version from five to three items and adapted the wording from referring to 'others' into the partner or one of the parents.
  Hofmann, S. G., Carpenter, J. K., & Curtiss, J. (2016). Interpersonal Emotion Regulation Questionnaire (IERQ): Scale development and psychometric characteristics. Cognitive Therapy and Research, 40(3), 341-356. https://doi.org/10.1007/s10608-016-9756-2
Adolescents quality of life (KIDSCREEN-10) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Increase in quality of life of adolescents (parents and adolescent will report about adolescent). Quality of life in terms of physical, mental, and social well-being will be determined by both the official parental and adolescent versions of the KIDSCREEN-10 (Ravens-Sieberer, 2006).
  Ravens-Sieberer, U. The Kidscreen Questionnaires: Quality of Life Questionnaires for Children and Adolescents; handbook; Pabst Science Publ.: Lengerich, Germany, 2006.
Perceived ARE from parent to adolescent (BARE-6) | Change from baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Increase in the accessibility and responsiveness of partners and parents (partners will report about their partner and adolescents and parents about the parent). Accessibility and responsiveness to the partner's and adolescent's needs will be assessed with the 6 item Brief Accessibility, Responsiveness and Engagement scale (BARE: Sandberg et al., 2012).
  Sandberg, J. G., Busby, D. M., Johnson, S. M., & Yoshida, K. (2012). The Brief Accessibility, Responsiveness, and Engagement (BARE) Scale: A tool for measuring attachment behavior in couple relationships. Family Process, 51(4), 512-526. https://doi.org/10.1111/j.1545-5300.2012.01422.x

OTHER OUTCOMES:
Attachment | baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Attachment (partners will report about their relationship with the partner, adolescents about the relationship with the parent). Attachment will be assessed with the Experiences in Close Relationships -Relationship Structures questionnaire in the official partner and parent-adolescent versions (ECR-RS; Fraley et al., 2011). Its nine items measure Anxiety about Rejection and Avoidance of Intimacy.
  Fraley, R. C., Heffernan, M. E., Vicary, A. M., & Brumbaugh, C. C. (2011). The experiences in close relationships-Relationship Structures Questionnaire: A method for assessing attachment orientations across relationships. Psychological assessment, 23(3), 615. https://doi.org/10.1037/a0022898
Emotional clarity (understanding own emotions) | baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Emotional Clarity (parent and adolescents will report about themselves). Emotional clarity will be measured with 5 items of the Difficulties in Emotion Regulation Scale (DERS; Roemer & Gratz, 2003). It measures Clarity, or understanding of own emotions.
Validation of emotions | baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Validation of emotions (parents and adolescent report about the parent). Validation of the adolescent by the parent will be measured with the Interpersonal Regulation Interaction Scale (IRIS; Swerdlow & Johnson, 2022). We shortened the original version from ten to five items and referred to one of the parents.
  Swerdlow, B. A., & Johnson, S. L. (2022). The Interpersonal Regulation Interaction Scale (IRIS): A multistudy investigation of receivers' retrospective evaluations of interpersonal emotion regulation interactions. Emotion, 22(6), 1119-1136. https://doi.org/10.1037/emo0000927
Apologizing and repair | baseline (pre-waiting, week 0) to post-intervention (week 5) and follow-up (week 13)
  Apologizing (parents and adolescent report about the parent). Apologizing of the parent to the adolescent will be measured with a self-constructed questionnaire based on the Proclivity to Apologize measure (PAM; Howell et al., 2011) and questions formulated by Bachman and Guerrero (2006).
  Bachman, G. F., & Guerrero, L. K. (2006). Fogiveness, Apology, and Communicative Responses to Hurtful Events. Communication Reports, 19(1-2), 45-56. https://doi.org/10.1080/08934210600586357
  Howell, A. J., Dopko, R. L., Turowski, J. B., & Buro, K. (2011). The disposition to apologize. Personality and Individual Differences, 51(4), 509-514. https://doi.org/10.1016/j.paid.2011.05.009
Observation of secure base behavior | one-time measurement at parent-adolescent session (week 4)
  Secure attachment behavior during the parent-adolescent session aiming at restoring the secure bond between parents and adolescent will be scored with the Secure Base Scoring Scale (Crowell et al., 2002), an observation instrument, based on the audio recording of this specific session. It contains three subscales: Availability, Sensitivity, and Responsiveness.
  Crowell, J. A., Treboux, D., Gao, Y., Fyffe, C., Pan, H., & Waters, E. (2002). Assessing secure base behavior in adulthood: Development of a measure, links to adult attachment representations and relations to couples' communication and reports of relationships. Developmental Psychology, 38(5), 679-693. https://doi.org/10.1037/0012-1649.38.5.679

CONTACTS AND LOCATIONS:
Overall Officials: Henk Jan Conradi, Doctor of Philosophy, Principal Investigator — University of Amsterdam
Locations (5):
- Netherlands (5):
  - Connected Together, Almere Stad
  - Molemann Mental Health, Almere Stad
  - Twig Clinics B.V., Bilthoven
  - Molemann Mental Health, Hilversum
  - Twig Clinics B.V., Woerden

IPD SHARING:
Plan to Share IPD: No
Currently decided that individual participant data (IPD) will not be shared due to the sensitive nature of the data, which involves minors and families in a clinical setting. Ensuring participant confidentiality is a priority, and current infrastructure does not support secure sharing of these data. Future data sharing may be considered if appropriate anonymization and data use agreements can be established.